CLINICAL TRIAL: NCT01229332
Title: A Phase I/II, Single-center, Randomized, Cross-over, Double-blind, Placebo-controlled Study Evaluating Safety, Tolerability and Pharmacokinetic Profile of Levodopa Following Administration of Subcutaneous Continuously-delivered Carbidopa Solution (ND0611) on the Top of Different Oral Dosage Forms of Levodopa/Carbidopa in Levodopa-treated Parkinson's Disease Patients With Motor Fluctuations
Brief Title: A Safety, Tolerability and Pharmacokinetic Study of ND0611 on the Top of Different Oral Dosage Forms of Levodopa/Carbidopa in Parkinson's Disease Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ND0611/002
Record Dates: First submitted 2010-10-03; First posted 2010-10-27 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Parkinson's Disease
Keywords: Motor fluctuations levodopa pharmacokinetics carbidopa solution continuous
MeSH Terms: conditions — Parkinson Disease | interventions — Sodium Chloride; Carbidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Carbidopa (Placebo Comparator)
  Interventions: Drug: Carbidopa
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — Continuous 24 h administration
  Arms: Placebo
Drug: Carbidopa — Continuous 24 h administration
  Arms: Carbidopa

SUMMARY:
A cross-over study, where ND0611 or placebo will be tested on top of 3 different LD/CD dosage forms. Safety and tolerability, pharmacokinetic profile of levodopa and carbidopa and the potential clinical effect of ND0611 will be explored in subjects with PD and motor fluctuations.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with idiopathic Parkinson's disease
2. Subjects must experience motor fluctuations associated with LD/CD dosing
3. Modified Hoehn and Yahr stage < 5
4. Subjects must be taking optimized and stable levodopa/dopa decarboxylase inhibitor therapy
5. Women must be postmenopausal, surgically sterilized, or using adequate birth control. Women of childbearing potential must have a negative pregnancy test (serum beta-HCG) at screening.
6. Subjects must be age 30 or older.
7. Subjects must be willing and able to give informed consent.

Exclusion Criteria:

1. Subjects with a clinically significant or unstable medical or surgical condition
2. Subjects with clinically significant psychiatric illness.
3. Pre-menopausal women, not using birth control method.
4. Subjects who have taken experimental medications within 60 days prior to baseline.
5. Subject who have undergone a neurosurgical intervention for Parkinson's disease (e.g., pallidotomy, thalamotomy, transplantation and deep brain stimulation).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence and frequency of adverse events, withdrawal rate | Up to 2 days
  1. Incidence and frequency of adverse events, of dopaminergic adverse events 2. Adverse events reporting related to the ND0611 Omnipod® application, Draize score 2. Withdrawal rates and discontinuations due to adverse events

SECONDARY OUTCOMES:
Half life (t½ ), Cmax, Tmax and AUC of levodopa and carbidopa in the plasma | Up to 2 days
  Pharmacokinetic profile of plasma LD and CD: Half life (t½ ), Cmax, Tmax and AUC
Half life (t½ ), Cmax, Tmax and AUC of levodopa and carbidopa in the plasma | Up to 2 days
  Pharmacokinetics profile of plasma LD and CD: Half life (t½ ), Cmax, Tmax and AUC

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel